CLINICAL TRIAL: NCT05442073
Title: Effect of Initial Empirical Positive End-Expiratory Pressure (PEEP) Setting on the Esophageal Pressure-guided PEEP Titration in Acute Respiratory Distress Syndrome
Brief Title: Effect of Initial Empirical PEEP Setting on the Esophageal Pressure-guided PEEP Titration in ARDS
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-2458
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: ARDS, Human; PEEP, Occult; Esophageal and Pleural Pressure
MeSH Terms: conditions — Respiratory Distress Syndrome; Positive-Pressure Respiration, Intrinsic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type I: ΔPes≥30%ΔPEEP
  Interventions: Other: PEEP adjustment
- Type II: ΔPes<30%ΔPEEP
  Interventions: Other: PEEP adjustment

INTERVENTIONS:
Other: PEEP adjustment — adjusting PEEP about 3-5cmH2O (increase or decrease)

SUMMARY:
Esophageal manometry was used as surrogate of pleural pressure to titrate positive end-expiratory pressure (PEEP) in ARDS patients. However, Absolute values of esophageal pressure (Pes) could be affected by the PEEP setting. In moderate to severe ARDS patients, the end-expiratory Pes changed differently with PEEP adjustment. and the esophageal phenotypes could be divided into type I and type II. with Type I （ΔPes≥30%ΔPEEP）and Type II（ΔPes<30%ΔPEEP）.

ELIGIBILITY:
Inclusion Criteria:

- aged over 18 all the moderate to severe ARDS patients invasive mechanical ventilation

Exclusion Criteria:

* aged<18 contraindication to esophageal catheter

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients all the moderate to severe ARDS with P/F<200 no contraindication to esophageal catheter
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
the changes of esophageal pressure during the PEEP titration | March 1st to May 31st, 2022

CONTACTS AND LOCATIONS:
Overall Officials: Shuyang Zhang, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No